CLINICAL TRIAL: NCT02286960
Title: Investigation of the Role of Steroids in Enhancing Voice Therapy Outcomes
Acronym: AAO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-00096
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid (Active Comparator): Prednizone pills. 4 day course 2 x 20mg per day.
  Interventions: Drug: Steroid
- Placebo (Placebo Comparator): Lactose Pills. 4 day course 2 x 20mg per day.
  Interventions: Dietary Supplement: Lactose Pills

INTERVENTIONS:
Drug: Steroid — A short 4 day course is administered to the first group of patients with voice disorders before the initiation of voice therapy.
  Other Names: Prednizone
  Arms: Steroid
Dietary Supplement: Lactose Pills — 4 day course 2 x 20mg per da
  Arms: Placebo

SUMMARY:
Despite the considerable use of oral steroids in the regular management of benign vocal fold lesions there is little evidence base in the literature. This study will investigate the efficacy of oral steroids for the treatment of vocal fold lesions in a controlled manner. The specific aim of this study is to determine the effectiveness of of a short course of oral steroids prior to behavioral voice therapy in patients with benign, phonotraumatic vocal fold lesions. Enrolled subjects will be randomized using a random numbers table to either receive oral steroids or no steroids prior to the initiation of voice therapy. The therapist and individuals involved in the collection and analysis of data will be blinded as to whether the subject received drug. Prior to initiation of therapy subjects will be asked to return for an interval evaluation during which they undergo videostroboscopy and voice evaluation. Subjects will enter then the voice therapy phase . After an initial evaluation to determine the best mode of therapy they will receive a behavioral voice therapy course, which includes a range of behavioral modifications and motor learning techniques, along with lifestyle measures. In all these phases acoustic and aerodynamic measurements will be collected as well as audio-visual material from the videostroboscopic exams. The investigators hypothesize that oral steroids will lead to a reduction in lesion size, which will substantially aid in the delivery and incorporation of voice therapy techniques, contributing to the improvement of overall laryngeal biomechanics and providing an ideal starting point for behavioral voice therapy.

DETAILED DESCRIPTION:
The study will investigate the potential added advantage of the use of steroids in patients undergoing voice therapy. Enrolled subjects will be randomized using a random numbers table to either receive oral steroids or no steroids prior to the initiation of voice therapy. The therapist and individuals involved in the collection and analysis of data will be blinded as to whether the subject received drug. Prior to initiation of therapy subjects will be asked to return for an interval evaluation during which they undergo videostroboscopy and voice evaluation. Subjects will enter then the voice therapy phase . After an initial evaluation to determine the best mode of therapy they will receive a behavioral voice therapy course, which includes a range of behavioral modifications and motor learning techniques, along with lifestyle measures. In all these phases acoustic and aerodynamic measurements will be collected as well as audio-visual material from the videostroboscopic exams. The measurements that will be collected in all these phases are the Voice Handicap Index (VHI)-10 , the noise to harmonic ratio H/N, the fundamental frequency Fo, The transglottic airflow and subglottic pressure. The investigators hypothesize that oral steroids will lead to a reduction in lesion size, which will substantially aid in the delivery and incorporation of voice therapy techniques, contributing to the improvement of overall laryngeal biomechanics and providing an ideal starting point for behavioral voice therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 males and females
* Presence of phonotraumatic lesion deemed to be etiologic for the complaint of dysphonia
* Voice therapy deemed to be the primary (or at least initial) treatment to address the dysphonia.
* Willingness to be an active participant in voice therapy.

Exclusion Criteria:

* Use of any glucocorticoids (oral, inhaled, or intravenous) within 3 months of the initial evaluation
* Known allergy or hypersensitivity to oral steroids
* Active infection
* Diabetes Mellitus
* Prior history of radiation to the neck
* Recent myocardial infarction
* Recent gastrointestinal surgery with bowel anastamosis (3 months)
* Active peptic ulcer
* Pregnancy
* Severe depression or history of psycosis
* History of recent laryngeal surgery (within 12 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Amin, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Steroid | Placebo
Started | 19 | 17
Completed | 16 | 14
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: A total of 6 patients were lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) Score From Baseline to 2 Months
Description: Data will be collected via measurement of the hatchmark on the 100mm line for each variable (e.g. 72/100). The higher the score, the higher the deviancy. The final score is the average of scores from each variable.
Time Frame: pre-treatment/baseline to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 14 | 13
score on a scale | 0.72 (0.21) | 0.65 (0.14)

2. Secondary Outcome: Change in Lesion Size From Baseline to 2 Months
Description: Still images of the glottis will be obtained from the video such that the vocal folds are captured in an open position (at least 40 degrees at the anterior commissure). Image J software (NIH) will then be used to outline the lesion and measure the length of the ipsilateral vocal fold.
Time Frame: pre-treatment/baseline to 2 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 14 | 13
mm | -0.4694 (0.5494) | 0.2788 (0.3026)

3. Secondary Outcome: Change in Voice Handicap Index (VHI) Scores From Baseline to 2 Months.
Description: A change in VHI scores from pre-treatment to following treatment.
  Scores can range from 0-120:
  0-30: Mild Minimal amount of handicap 31-60: Moderate Often seen in patients with vocal nodules, polyps, or cysts 60-120: Severe Often seen
Time Frame: Pre-treatment/baseline to following treatment/2 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 14 | 13
score on a scale | 0.35 [-.2 to .9] | 0.40 [.15 to .95]

4. Secondary Outcome: Number of Participants That Showed Improved (Lower) Average Decibels (db) Output.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 14 | 13
Participants | 14 | 13

ADVERSE EVENTS:
Time Frame: 2 Months
Arm/Group | Steroid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02286960/Prot_SAP_000.pdf